CLINICAL TRIAL: NCT02496858
Title: Clinical and Genetic Characteristics of Coronary Artery Disease in Chinese Young Adults
Acronym: GRAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Dr., Shanghai Zhongshan Hospital
Other Study IDs: ZS-CV-2015
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Young Patient; Genetic Characteristics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 samples of EDTA blood (2ml glass) and 1 sample of serum (2ml glass) will be retained in a biobank.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Early-onset CAD: The anticipated 2000 young CAD patients who aged ≤45years undergoing coronary angiography will be recruited in the prospective cohort. Medical history and risk-factor information were obtained by interviewing patients and by abstracting information from medical records.
- Late-onset CAD: The anticipated 2000 old CAD patients aged≥65years undergoing coronary angiography will be recruited in the prospective cohort. Medical history and risk-factor information were obtained by interviewing patients and by abstracting information from medical records.
- Age-matched controls: The anticipated 2000 control subjects without obvious coronary stenosis aged≤45years or ≥65years will be recruited in the prospective cohort. Medical history and risk-factor information were obtained by interviewing patients and by abstracting information from medical records.

SUMMARY:
The aim of this study is to identify genetic loci,or gene variations contributing to the development of coronary artery disease (CAD) in Chinese young adults. Investigators will compare coronary angiogram results to genetic findings within young CAD patients.

DETAILED DESCRIPTION:
During last 10 years, the rise in coronary artery disease (CAD) prevalence in Chinese young adults is observed and percutaneous coronary intervention (PCI) is generally considered to be low operative risk in these young patients. Genome-wide association studies have identified a considerable number of common genetic variants related to CAD. However, the extent to which these genetic variants are related to the future cardiovascular events, the prevalence, extent, severity, and prognosis of young patients with CAD is not clear.

The aim of this study is to investigate the genetic loci, or gene variations contributing to the development and prognosis of CAD in Chinese young adult. Investigators will compare the angiogram results to genetic findings first in patients with different stages of CAD. Then, investigators will collect patients from hospital discharge registry, and compare long-term outcome as well as on operative details in different gene groups.

The results of the study provide a possibility to develop a gene test to recognize patients at risk at its early stage, and needing for preventive medicine.

ELIGIBILITY:
Inclusion criteria:

1. premature CAD, includes patients who aged ≥ 18 and ≤ 45 years , and with at least one main coronary artery stenosis ≥ 50% confirmed by coronary angiography, involving left main coronary artery, left anterior descending branch, left circumflex branch or right coronary artery, and manifested as occult CAD, stable CAD, unstable angina pectoris, non-ST segment elevated myocardial infarction and ST segment elevated myocardial infarction;
2. mature CAD, refers to patients who aged ≥ 65 years and meat the same CAD diagnostic criteria as above;
3. age matched individuals who had coronary arteries without obvious stenosis.

Exclusion criteria:

1. severely sick with limited life-expectancy < 1 year;
2. patients with malignancies;
3. pregnant or planning for pregnancy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged ≤45 years diagnosed with CAD by coronary angiography will be collected from multiple institutions.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Number of cardiac death | 36 months
  Any death from cardiac conditions
Number of patients developing myocardial infarction | 36 months
  Any case of acute myocardial infarction which meet the Criteria according to current guidelines.
Number of patients developing stroke | 36 months
  Any events of ishcemic stroke, TIA or hemorrhagic stroke
Number of participants undergoing unscheduled repeat revascularization of target or non-target vessel | 36 months
  Any unshceduled percutaneous coronary intervention or coronary artery bypass grafting after primary revascularization

SECONDARY OUTCOMES:
Number of stent thrombosis, bleeding、non-cardiac death and all-cause death. | 36 months
  Composite of stent thrombosis, bleeding、non-cardiac death and all-cause death.

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Zhuhai Hospital of Guangdong Provincial People's Hospital, Zhuhai, Guangdong
  - The First Affiliated Hospital of Guangxi University of Traditional Chinese Medicine, Nanning, Guangxi
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - The second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuxi Third People's Hospital, Wuxi, Jiangsu
  - Xuzhou Fourth People's Hospital, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The second Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Central Hospital of Jiading District, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai, Shanghai Municipality
  - Central Hospital of Yangpu District, Shanghai, Shanghai Municipality
  - Changhai Hospital of Second Military Medical University of Chinese PLA, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai chest hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Shidong Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Yueyang hospital, Shanghai, Shanghai Municipality
  - Shanxi cardiovascular hospital, Taiyuan, Shanxi
  - Taiyuan central hospital, Taiyuan, Shanxi
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Karamay Central Hospital, Karamay, Xinjiang
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhenjiang First People's Hospital, Hangzhou, Zhenjiang

REFERENCES:
- [Derived] Wu R, Su Y, Liao J, Shen J, Ma Y, Gao W, Dong Z, Dai Y, Yao K, Ge J. Exome Sequencing Identified Susceptible Genes for High Residual Risks in Early-Onset Coronary Atherosclerotic Disease. Clin Cardiol. 2024 Dec;47(12):e70066. doi: 10.1002/clc.70066. PMID 39673281